CLINICAL TRIAL: NCT05254327
Title: A Randomized Phase 2 Trial of the Efficacy and Safety of Short and Long Course Radiation Therapy With and Without BMX-001 as Part of Total Neoadjuvant Therapy in Patients With Newly Diagnosed Locally Advanced Rectal Adenocarcinoma
Brief Title: Trial of the Efficacy and Safety of Short and Long Course Radiation Therapy With/Without BMX-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: BioMimetix JV, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0012-22-FB; BMX-RAC-001 (Other: BioMimetix JV, LLC)
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer
Keywords: Radiation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Lab performing PK sample analysis will be blinded to the subjects and relationship of specimens to treatment with BMX-001
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Experimental): Short Chemo-Radiation Therapy (SCRT) + BMX-001
  Interventions: Drug: BMX-001
- Arm B (No Intervention): Short Chemo-Radiation Therapy (SCRT)
- Arm C (Experimental): Long Course Chemo-Radiation Therapy (LCCRT) + BMX-001
  Interventions: Drug: BMX-001
- Arm D (No Intervention): Long Course Chemo-Radiation Therapy (LCCRT)

INTERVENTIONS:
Drug: BMX-001 — Loading dose of 28 mg per subject, followed by maintenance doses of 14 mg per subject twice per week.
  Arms: Arm A; Arm C

SUMMARY:
In this Phase 2 study, we will conduct an efficacy and safety study of the combination of investigational drug BMX-001, with short-course radiotherapy (SCRT) or long-course chemoradiotherapy (LCCRT) as part of total neoadjuvant therapy in newly diagnosed rectal adenocarcinoma (RAC) patients.

DETAILED DESCRIPTION:
In this trial, we will enroll patients in two cohorts:

Cohort 1: A 6 patient safety lead-in for patients receiving capecitabine prior to beginning a randomized trial for the Long Course Chemo-radiation (LCCRT) cohort. There will be trial stopping rules to review safety and PK data prior to initiating the randomized trial of patients receiving LCCRT.

Cohort 2: The Randomized Short Course Radiation (SCRT) cohort.

Cohort 1 and 2 will begin enrolling concurrently. Cohort 1 will have a safety lead-in of patients receiving LCCRT (with capecitabine). Cohort 2 will begin with the randomized study of patients receiving SCRT, while the LCCRT cohort is going through the safety lead-in portion.

There are stopping rules for the LCCRT cohort 1 pending PK analysis as well as an AE review from the treatment period plus 1 week post BMX-001 treatment for the 6 patients prior to moving on with the randomized portion of the study for the LCCRT cohort. All patients in the safety lead-in portion of the trial will receive BMX-001 (A loading dose of 28 mg/subject followed by maintenance doses of 14 mg/subject twice a week) with either SCRT or LCCRT. Patients will receive 3 cycles of FOLFOX or 2 cycles of CAPOX and then be assigned to SCRT or LCCRT prior to randomization. Patients will be randomized (stratified by gender) to BMX-001 or no BMX-001. The randomized trial in each cohort will involve SCRT or LCCRT with or without BMX-001. After conclusion of radiation, patients will then receive 6 more cycles of FOLFOX or 4 more cycles of CAPOX. Skin, GI, and GU symptoms will be measured on the day of screening, before and after RT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed locally advanced rectal adenocarcinoma who will be receiving total neoadjuvant therapy regimen with curative intent.
2. AJCC stage II to III rectal adenocarcinoma that will require total neoadjuvant therapy.
3. Adult, age > or equal to 18 years (for Nebraska, age of consent is ≥19 years old)
4. ECOG Performance Status 0-2
5. Hemoglobin ≥ 9.0 g/dl, ANC ≥ 1,500 /dl, platelets ≥ 100,000 /dl (The use of transfusion or other intervention to achieve Hgb > 9.0 g/dl is acceptable)
6. Serum SGOT and bilirubin ≤ 1.5 times upper limit of normal
7. Adequate renal function defined as follows:

1)Serum creatinine < 1.5 mg/dl within 2 weeks prior to enrollment or 2)Creatinine clearance (CC) ≥ 50 ml/min within 2 weeks prior to enrollment determined by 24-hour collection or estimated by Cockcroft-Gault formula: CCr male = [(140 - age) x (wt in kg)]/[(Serum Cr mg/dl) x (72)], CCr female = 0.85 x (CrCl male) 8. Signed, written informed consent prior to completing any study specific procedures 9. Negative pregnancy test for women of child-bearing potential at the time of screening 10. Women of childbearing potential and male participants must agree to use two forms of a medically effective means of birth control throughout their participation in the treatment phase of the study and until 12 months following the last study treatment 11. Chest/Abdominal/Pelvic (CAP) CT/ pelvic MRI done within 8 weeks prior to randomization.

Exclusion Criteria:

1. Breast-feeding or pregnant
2. Active infection requiring IV antibiotics 7 days before enrollment
3. Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ, basal cell or carcinoma of the skin, invasive cancers with a 5-year disease-free interval, resected cancer of the bladder or low-grade (Gleason 6 or less) prostate cancer
4. Prior history of rectal adenocarcinoma (RAC)
5. Prior history of pelvic radiotherapy for any other type of malignancy
6. Known hypersensitivity or contraindication to any agent in FOLFOX or CAPOX regimen.
7. Because corticosteroids are anti-inflammatory and could interrupt oxidative stress, patients will be excluded unless they are on stable or decreasing corticosteroids dose at the time of randomization.

   BMX-001 Specific Exclusion Criteria (Subjects meeting any of the following criteria are ineligible for study entry)
8. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg)
9. Active or history of postural hypotension and autonomic dysfunction within the past year
10. Known hypersensitivity to BMX-001
11. Clinically significant (i.e. active) cardiovascular disease or cerebrovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
12. History or evidence upon physical/neurological examination of central nervous system disease (e.g. seizures) unrelated to cancer unless adequately controlled by medication or potentially interfering with protocol treatment
13. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment
14. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds (ms) (CTCAE grade 1) using the specific/usual choice by clinical center for correction factor.
15. A history of additional risk factors for Torsades de Pointes (TdP) (e.g., congestive heart failure, hypokalemia, known family history of Long QT Syndrome).

Note: Inclusion of Women and Minorities Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy of BMX-001 as measured by Grade 3 and above associated with gastrointestinal Toxicities | Three weeks (During and 2 weeks after RT)
  Grade 3 and above radiation-associated gastrointestinal, genitourinary, skin and hematologic toxicity (SCRT or LCCRT) including frequency, severity and duration of rectal bleeding, rectal pain, diarrhea, dysuria, hematuria, urinary frequency, radiation dermatitis and thrombocytopenia
Efficacy of BMX-001 as measured by Grade 3 and above associated with genitourinary Toxicities | Three weeks (During and 2 weeks after RT)
  Grade 3 and above radiation-associated gastrointestinal, genitourinary, skin and hematologic toxicity (SCRT or LCCRT) including frequency, severity and duration of rectal bleeding, rectal pain, diarrhea, dysuria, hematuria, urinary frequency, radiation dermatitis and thrombocytopenia
Efficacy of BMX-001 as measured by Grade 3 and above associated with skin Toxicities | Three weeks (During and 2 weeks after RT)
  Grade 3 and above radiation-associated gastrointestinal, genitourinary, skin and hematologic toxicity (SCRT or LCCRT) including frequency, severity and duration of rectal bleeding, rectal pain, diarrhea, dysuria, hematuria, urinary frequency, radiation dermatitis and thrombocytopenia
Efficacy of BMX-001 as measured by Grade 3 and above associated with hematologic Toxicities | Three weeks (During and 2 weeks after RT)
  Grade 3 and above radiation-associated gastrointestinal, genitourinary, skin and hematologic toxicity (SCRT or LCCRT) including frequency, severity and duration of rectal bleeding, rectal pain, diarrhea, dysuria, hematuria, urinary frequency, radiation dermatitis and thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Chi Lin, MD, PhD, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - Markey Cancer Center, Lexington, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - UT Health San Antonio MD Anderson Cancer Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No